CLINICAL TRIAL: NCT02436382
Title: The Impact of Ambient Operative Room Temperature on Neonatal and Maternal Hypothermia
Brief Title: Hypothermia and the Effect of Ambient Temperature
Acronym: HEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Elaine Duryea, Fellow Physician, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU 122014-046
Record Dates: First submitted 2015-01-30; First posted 2015-05-06 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Hypothermia
MeSH Terms: conditions — Hypothermia | interventions — Temperature

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ambient Temperature of 67F (No Intervention): These patients will have an operating room temperature of 67F for cesarean delivery, the standard of care at our institution.
- Ambient Temperature of 73F (Active Comparator): These patient will have an operating room temperature of 73F for cesarean delivery, a temperature more consistent with WHO recommendations.
  Interventions: Other: change in temperature

INTERVENTIONS:
Other: change in temperature — increase in ambient room temperature
  Arms: Ambient Temperature of 73F

SUMMARY:
Neonatal hypothermia is associated with increased risk of mortality as well as multiple morbidities. The investigators objective is to determine if an increase in ambient operative room temperature decreases the rate of hypothermia. Operating room temperature will be randomized to the current institutional standard (67°F) or a temperature of 73°F on a weekly basis for a period of six months.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women and their neonates undergoing cesarean delivery by the Parkland Hospital Obstetrics Service on the Labor and Delivery "West" Unit (operating rooms 1, 2, 3, and 5) during the study period.

Exclusion Criteria:

* Subjects will be excluded from the study if cesarean delivery is planned but a precipitous vaginal delivery occurs, intrauterine fetal demise has been diagnosed prior to start of surgery, the neonate is noted to have a major congenital anomaly, resuscitative efforts are not performed ("comfort care only" provided), or a neonatal temperature is not available.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 846 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
neonatal hypothermia | up to 2 hours following delivery
  a core temperature of less than 36.5C

SECONDARY OUTCOMES:
maternal hypothermia | up to 10 hours following delivery
  an oral temperature of less than 36.5C

OTHER OUTCOMES:
neonatal hypoglycemia | up to 8 hours following delivery
  hypoglycemia requiring treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Parkland Memorial Hospital, Dallas, Texas, United States